CLINICAL TRIAL: NCT03451162
Title: A Phase I, Open-Label Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Escalating Doses of DHES0815A in Patients With HER2-Positive Breast Cancer
Brief Title: Safety, Tolerability, and Pharmacokinetic (PK) Study of DHES0815A in Participants With Human Epidermal Growth Factor Receptor (HER)2-Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO39869
Record Dates: First submitted 2018-02-16; First posted 2018-03-01 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — DHES0815A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort: DHES0815A (Experimental): Participants will receive DHES0815A in escalating doses in the dose-escalation cohort of the study. Participants will receive additional infusions of DHES0815A on Day 1 of subsequent cycles provided that they meet the protocol specified criteria for acceptable toxicity and ongoing clinical benefit.
  Interventions: Drug: DHES0815A
- Dose Expansion Cohort: DHES0815A (Experimental): Participants will be treated at or below the Maximum Tolerated Dose (MTD) of DHES0815A (based on the review of the totality of the data) to obtain additional safety, tolerability, PK, and anti-tumor activity data.
  Interventions: Drug: DHES0815A

INTERVENTIONS:
Drug: DHES0815A — DHES0815A will be administered via intravenous (IV) infusion on Day 1 of each 21-day cycle.

SUMMARY:
This first-in-human, Phase 1, open-label, multicenter, dose-escalation study will evaluate the safety, tolerability, and PK of DHES0815A as a single agent in participants with advanced and/or metastatic HER2-positive breast cancer for whom established treatment has proven ineffective or intolerable or is unavailable. The study may include a dose-expansion cohort (based on an ongoing assessment of the totality of data obtained in this study) to further assess safety, tolerability, PK, and preliminary anti-tumor activity.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease by RECIST v1.1 with at least one measurable target lesion
* Locally advanced or metastatic HER2-positive breast cancer that has relapsed or is refractory to established therapies
* Adequate hematologic and end-organ function
* For dose-expansion cohort only: no more than two prior systemic chemotherapy-containing regimens in the advanced/metastatic setting (excluding trastuzumab emtansine, which is considered a targeted cytotoxic agent)

Key Exclusion Criteria:

* Treatment with chemotherapy, hormonal therapy (except hormone replacement therapy, oral contraceptives), immunotherapy, biologic therapy, radiation therapy (except palliative radiation to bony metastases), or herbal therapy as cancer therapy within 4 weeks prior to initiation of DHES0815A
* History of exposure to the protocol specified doses of anthracyclines
* Pregnancy, lactation, or breastfeeding
* Major surgical procedure within 4 weeks prior to Day 1
* Evidence of a significant uncontrolled concomitant disease of the nervous system, pulmonary, autoimmune, renal, hepatic, endocrine, or gastrointestinal disorders; or a serious non-healing wound or fracture
* Known active bacterial, viral, fungal, mycobacterial, or other infection
* Clinically significant history of liver disease, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* Untreated or active central nervous system (CNS) metastases
* Cardiopulmonary dysfunction, including inadequate left ventricular ejection function at baseline, less than 50% by either echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* QT interval corrected through use of Fridericia's formula (QTcF) > 470 milliseconds (ms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lewis GD, Li G, Guo J, Yu SF, Fields CT, Lee G, Zhang D, Dragovich PS, Pillow T, Wei B, Sadowsky J, Leipold D, Wilson T, Kamath A, Mamounas M, Lee MV, Saad O, Choeurng V, Ungewickell A, Monemi S, Crocker L, Kalinsky K, Modi S, Jung KH, Hamilton E, LoRusso P, Krop I, Schutten MM, Commerford R, Sliwkowski MX, Cho E. The HER2-directed antibody-drug conjugate DHES0815A in advanced and/or metastatic breast cancer: preclinical characterization and phase 1 trial results. Nat Commun. 2024 Jan 11;15(1):466. doi: 10.1038/s41467-023-44533-z. PMID 38212321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 5 investigative sites in Republic of Korea and United States from 17 April 2018 to 16 July 2021.
Pre-assignment Details: No participants were enrolled in the Dose Expansion Cohort.
Groups:
- Dose Escalation Cohort: DHES0815A 0.6 mg/kg: Participants received DHES0815A 0.6 milligrams per kilograms (mg/kg) as an intravenous (IV) infusion, every three weeks (Q3W) on Day 1 of each 21-day cycle.
- Dose Escalation Cohort: DHES0815A 1.2 mg/kg: Participants received DHES0815A 1.2 mg/kg as an IV infusion, Q3W on Day 1 of each 21-day cycle.
- Dose Escalation Cohort: DHES0815A 2.4 mg/kg: Participants received DHES0815A 2.4 mg/kg as an IV infusion, Q3W on Day 1 of each 21-day cycle.
- Dose Escalation Cohort: DHES0815A 4 mg/kg: Participants received DHES0815A 4 mg/kg as an IV infusion, Q3W on Day 1 of each 21-day cycle up to Cycle 3. Due to toxicities observed in participants after Cycle 3, dosing was capped at 2.4 mg/kg and the participants received DHES0815A at a dose of 2.4 mg/kg as an IV infusion, Q3W from Cycle 4, on Day 1 of each 21-day cycle.
- Dose Escalation Cohort: DHES0815A 6 mg/kg: Participants received DHES0815A 6 mg/kg as IV infusion, Q3W on Day 1 of each 21-day cycle. Due to toxicities observed in participants after 3 cycles of DHES0815A 4 mg/kg, dosing was capped at 2.4 mg/kg and the participants received DHES0815A at a dose of 2.4 mg/kg as an IV infusion, Q3W from Cycle 4, on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Started | 3 | 3 | 3 | 3 | 2
Completed | 1 | 1 | 3 | 3 | 2
Not Completed | 2 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (6.1) | 58.3 (4.5) | 49.3 (8.3) | 48.3 (5.0) | 50.0 (15.6) | 54.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 2 | 14
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 2 | 3 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 2 | 2 | 1 | 2 | 2 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) With Severity Determined as Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Description: AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. SAE is any AE that is fatal, is life threatening, requires or prolongs inpatient hospitalization, results in persistent/significant disability/incapacity and is congenital anomaly/birth defect. Severity of AEs were graded per NCI CTCAE v4.0. Grade 1: Mild; asymptomatic/mild symptoms; clinical/diagnostic observations only; or intervention not indicated; Grade 2: Moderate; minimal, local/non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3: Severe/medically significant, but not immediately life-threatening: hospitalization/prolongation of hospitalization indicated; disabling/limiting self-care activities of daily living; Grade 4: Life-threatening consequences/urgent intervention indicated; Grade 5: Death related to AE.
Time Frame: From Day 1 to end of study (up to approximately 39 months)
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
Participants
  AEs | 3 | 3 | 3 | 3 | 2
  SAEs | 1 | 1 | 1 | 0 | 1
  Grade 1 AEs | 0 | 0 | 1 | 0 | 0
  Grade 2 AEs | 1 | 2 | 0 | 1 | 1
  Grade 3 AEs | 1 | 1 | 2 | 2 | 1
  Grade 4 AEs | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: DLT=any one events occurring during DLT assessment window: ≥15% decrease from baseline in left ventricular ejection fraction (LVEF)/≥10% decrease to <50% LVEF; Grade ≥ 3 non-hematologic toxicity; Grade ≥4 neutropenia (absolute neutrophil count <500 cells/microliters [μL]) lasting <7 days; Grade ≥3 febrile neutropenia; Grade ≥4 anemia; Grade ≥4 thrombocytopenia; Grade 3 thrombocytopenia associated with clinically significant bleeding; Any increase in hepatic transaminase (ALT or AST) >3*baseline in combination with either an increase in direct bilirubin >2*upper limit of normal/clinical jaundice, in absence of cholestasis/other contributory factors. NCI CTCAE v4.0. was used to grade these events.Grade1: Mild; asymptomatic/mild symptoms; clinical/diagnostic observations only; Grade2: Moderate; minimal, local/non-invasive intervention indicated;Grade3: Severe/medically significant, but not immediately life-threatening;Grade4: Life-threatening consequences/urgent intervention indicated.
Time Frame: From Day 1 up to Day 21
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Duration of Treatment
Description: Treatment duration was calculated from the first dose of study drug to the last dose of study drug administration.
Time Frame: From Day 1 up to last dose of study drug (up to approximately 39 months)
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
days | 64.0 [62 to 533] | 208.0 [85 to 960] | 43.0 [43 to 66] | 64.0 [64 to 127] | 43.0 [43 to 43]

4. Primary Outcome: Total Cumulative Dose
Time Frame: From Day 1 up to last dose of study drug (up to approximately 39 months)
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
milligrams (mg) | 882.33 (1355.91) | 2143.00 (2523.37) | 342.27 (157.78) | 1340.20 (586.56) | 548.80 (138.59)

5. Primary Outcome: Change From Baseline in LVEF as Assessed by Echocardiogram (ECHO) or Multiple-Gated Acquisition (MUGA) Scan
Description: LVEF is the fraction of blood (in percent) pumped out of the heart's left ventricular chamber with each heartbeat and is a measure of cardiac output for the heart. Baseline LVEF value and the change from baseline to the worst value in LVEF measurement were reported. LVEF was measured by ECHO or MUGA scan.
Time Frame: Baseline, end of Cycle 1, Days 15-21 of Cycles 2, 4, and 6, and every four cycles thereafter up to the study discontinuation visit (up to approximately 39 months)
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: percentage points of LVEF
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
percentage points of LVEF
  Baseline | 59.00 (3.61) | 63.33 (4.04) | 64.00 (9.54) | 59.67 (0.58) | 62.50 (3.54)
  Change From Baseline to Worst Value | 0.33 (4.04) | -1.67 (1.15) | -4.67 (7.77) | -1.33 (1.53) | -5.00 (0.00)

6. Secondary Outcome: Concentration of DHES0815A Total Antibody
Description: DHES0815A total antibody is one of three key pharmacokinetic analytes of DHES0815A.
Time Frame: Pre-dose and 30 minutes (min) post-dose on Day 1 Cycles 1-4; 4 hour (h) post-dose on Day 1 Cycle1; post-dose on Days 2, 3, 11, 17 Cycle 1; post-dose on Days 8 and 15 Cycles 1-4; study discontinuation visit (up to approx. 39 months) (Cycle length=21 days)
Population: Pharmacokinetics (PK) evaluable population included all enrolled participants who received at least one dose of study medication. Number analyzed is the number of participants with evaluable data at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
nanograms per milliliters (ng/mL)
  Cycle 1 Day1: Predose | NA (NA) — The data was not evaluable as the samples were below limit of quantification (BLQ). | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ.
  Cycle 1 Day 1: 30 min Postdose | 13100 (27.2) | 48700 (29.0) | 49200 (27.3) | 88600 (11.4) | 119000 (0.0)
  Cycle 1 Day 1: 4 h Postdose | 12200 (30.7) | 30500 (13.0) | 46900 (19.2) | 85900 (13.6) | 106000 (0.0)
  Cycle 1 Day 2 | 8460 (34.9) | 27000 (18.7) | 35500 (46.5) | 69100 (13.2) | 96800 (11.6)
  Cycle 1 Day 3: number analyzed (Participants) | 3 | 3 | 3 | 2 | 2
  Cycle 1 Day 3 | 6330 (37.1) | 22000 (14.5) | 26600 (52.3) | 59700 (9.7) | 81100 (15.8)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2
  Cycle 1 Day 8 | 625 (411.4) | 8120 (42.1) | 10700 (76.8) | 36000 (8.8) | 48000 (6.3)
  Cycle 1 Day 11: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
  Cycle 1 Day 11 | 225 (NA) — Values were less than reportable (LTR) for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 4870 (34.2) | 6840 (90.1) | 26000 (5.1) | 42100 (26.7)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 2 | 2
  Cycle 1 Day 15 | 64.8 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 2160 (69.1) | 2100 (135.7) | 22800 (0.3) | 31300 (27.7)
  Cycle 1 Day 17 | 50.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 1030 (190.3) | 981 (148.8) | 18800 (28.3) | 29700 (36.7)
  Cycle 2 Day 1: Predose | 50.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 66.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 50.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 10500 (46.2) | 19900 (27.3)
  Cycle 2 Day 1: 30 min Postdose | 11900 (29.6) | 33000 (28.8) | 30800 (101.0) | 97700 (15.8) | 85400 (62.2)
  Cycle 2 Day 8: number analyzed (Participants) | 3 | 3 | 2 | 3 | 1
  Cycle 2 Day 8 | 933 (165.1) | 9500 (11.1) | 10800 (46.2) | 44300 (8.5) | 80000 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.
  Cycle 2 Day 15: number analyzed (Participants) | 3 | 3 | 2 | 3 | 2
  Cycle 2 Day 15 | 50.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 2230 (37.2) | 1330 (78.7) | 27600 (12.9) | 31100 (123.0)
  Cycle 3 Day 1: Predose: number analyzed (Participants) | 3 | 3 | 1 | 3 | 0
  Cycle 3 Day 1: Predose | 50.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 50.00 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 50.0 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 18900 (38.9) |
  Cycle 3 Day 1: 30 min Postdose: number analyzed (Participants) | 3 | 3 | 1 | 3 | 0
  Cycle 3 Day 1: 30 min Postdose | 13600 (21.6) | 39300 (52.9) | 56900 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 119000 (14.1) |
  Cycle 3 Day 8: number analyzed (Participants) | 2 | 3 | 1 | 3 | 0
  Cycle 3 Day 8 | 765 (921.0) | 9740 (19.7) | 8720 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 51900 (20.0) |
  Cycle 3 Day 15: number analyzed (Participants) | 3 | 3 | 0 | 3 | 0
  Cycle 3 Day 15 | 50.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 2530 (66.3) |  | 30200 (24.7) |
  Cycle 4 Day 1: Predose: number analyzed (Participants) | 2 | 3 | 0 | 1 | 0
  Cycle 4 Day 1: Predose | 50.0 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 65.8 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. |  | 13800 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 1: 30 min Postdose: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 1: 30 min Postdose | 8750 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 32800 (16.8) |  | 83900 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 8: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 8 | 2130 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 11100 (23.5) |  | 24200 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 15 | 50.0 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 3000 (72.6) |  | 13500 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Study Drug Discontinuation Visit: number analyzed (Participants) | 2 | 2 | 3 | 2 | 1
  Study Drug Discontinuation Visit | 231 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 483 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 75.5 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 50.0 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 27800 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.

7. Secondary Outcome: Concentration of Plasma Conjugated Pyrrolo [2,1-c] [1,4] Benzodiazepine Monoamide (PDB-MA)
Description: Conjugated PDB-MA is one of three key pharmacokinetic analytes of DHES0815A.
Time Frame: as for outcome 6
Population: PK evaluable population included all enrolled participants who received at least one dose of study medication. Number analyzed is the number of participants with evaluable data at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
ng/mL
  Cycle 1 Day1: Predose | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ.
  Cycle 1 Day 1: 30 min Postdose | 90.5 (23.4) | 242 (11.4) | 381 (28.0) | 702 (3.8) | 864 (4.4)
  Cycle 1 Day 1: 4 h Postdose | 84.4 (28.9) | 234 (9.4) | 338 (31.0) | 666 (6.7) | 837 (4.6)
  Cycle 1 Day 2 | 55.6 (32.8) | 186 (7.6) | 234 (44.6) | 508 (8.0) | 693 (5.4)
  Cycle 1 Day 3: number analyzed (Participants) | 3 | 3 | 3 | 2 | 2
  Cycle 1 Day 3 | 38.2 (32.5) | 147 (8.1) | 183 (48.4) | 440 (1.4) | 577 (12.9)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2
  Cycle 1 Day 8 | 3.52 (394.8) | 53.8 (39.5) | 58.2 (69.4) | 225 (5.6) | 328 (5.2)
  Cycle 1 Day 11: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
  Cycle 1 Day 11 | 2.04 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 29.9 (33.7) | 33.0 (71.7) | 157 (6.4) | 259 (26.2)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 2 | 2
  Cycle 1 Day 15 | 0.947 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 11.6 (74.0) | 10.5 (122.9) | 118 (6.6) | 174 (28.4)
  Cycle 1 Day 17 | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 4.45 (313.1) | 4.40 (120.8) | 82.9 (29.5) | 160 (34.3)
  Cycle 2 Day 1: Predose | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 44.9 (59.5) | 90.6 (32.1)
  Cycle 2 Day 1: 30 min Postdose | 92.8 (14.7) | 247 (19.4) | 232 (92.5) | 760 (10.4) | 636 (53.8)
  Cycle 2 Day 8: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 2 Day 8 | 5.01 (182.3) | 59.5 (14.7) | 30.9 (183.6) | 283 (11.5) | 451 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.
  Cycle 2 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 2 Day 15 | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 11.5 (35.6) | 3.25 (224.3) | 135 (16.3) | 324 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.
  Cycle 3 Day 1: Predose: number analyzed (Participants) | 3 | 3 | 1 | 3 | 0
  Cycle 3 Day 1: Predose | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.750 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 76.3 (47.0) |
  Cycle 3 Day 1: 30 min Postdose: number analyzed (Participants) | 3 | 3 | 1 | 3 | 0
  Cycle 3 Day 1: 30 min Postdose | 100 (12.1) | 236 (17.5) | 381 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 803 (7.7) |
  Cycle 3 Day 8: number analyzed (Participants) | 2 | 3 | 1 | 3 | 0
  Cycle 3 Day 8 | 3.63 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 57.9 (16.5) | 61.6 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 294 (20.7) |
  Cycle 3 Day 15: number analyzed (Participants) | 3 | 3 | 0 | 3 | 0
  Cycle 3 Day 15 | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 12.1 (53.9) |  | 143 (30.8) |
  Cycle 4 Day 1: Predose: number analyzed (Participants) | 2 | 3 | 0 | 1 | 0
  Cycle 4 Day 1: Predose | 0.750 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.750 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. |  | 58.6 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 1: 30 min Postdose: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 1: 30 min Postdose | 112 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 244 (17.0) |  | 647 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 8: number analyzed (Participants) | 0 | 3 | 0 | 1 | 0
  Cycle 4 Day 8 |  | 55.8 (10.6) |  | 139 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0
  Cycle 4 Day 15 | 0.750 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 13.8 (70.4) |  |  |
  Study Drug Discontinuation Visit: number analyzed (Participants) | 1 | 2 | 3 | 0 | 0
  Study Drug Discontinuation Visit | 0.750 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 3.93 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 1.38 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. |  |

8. Secondary Outcome: Concentration of Plasma Unconjugated PDB-MA
Description: Plasma Unconjugated PDB-MA is one of three key pharmacokinetic analytes of DHES0815A.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
ng/mL
  Cycle 1 Day1: Predose | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ. | NA (NA) — The data was not evaluable as the samples were BLQ.
  Cycle 1 Day 1: 30 min Postdose | 0.107 (14.4) | 0.362 (40.9) | 0.497 (47.1) | 0.772 (9.1) | 1.05 (5.4)
  Cycle 1 Day 1: 4 h Postdose | 0.0770 (20.2) | 0.276 (16.9) | 0.328 (26.9) | 0.546 (21.4) | 0.985 (44.5)
  Cycle 1 Day 2 | 0.0634 (27.8) | 0.175 (2.9) | 0.223 (72.6) | 0.449 (43.9) | 0.577 (18.5)
  Cycle 1 Day 3: number analyzed (Participants) | 3 | 3 | 3 | 2 | 2
  Cycle 1 Day 3 | 0.0568 (31.8) | 0.130 (21.8) | 0.179 (40.2) | 0.252 (24.7) | 0.332 (14.5)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 2 | 3 | 3 | 2
  Cycle 1 Day 8 | 0.0300 (6.1) | 0.0800 (15.0) | 0.0927 (25.0) | 0.185 (32.4) | 0.163 (37.7)
  Cycle 1 Day 11: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
  Cycle 1 Day 11 | 0.0172 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0605 (16.8) | 0.0806 (15.2) | 0.146 (54.3) | 0.170 (43.2)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 2 | 2
  Cycle 1 Day 15 | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0405 (19.7) | 0.0490 (48.5) | 0.110 (47.6) | 0.103 (4.9)
  Cycle 1 Day 17 | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0337 (16.2) | 0.0389 (54.4) | 0.0896 (40.4) | 0.101 (37.4)
  Cycle 2 Day 1: Predose | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0178 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0836 (69.5) | 0.0991 (60.4)
  Cycle 2 Day 1: 30 min Postdose | 0.0969 (16.4) | 0.324 (29.7) | 0.321 (73.3) | 0.953 (17.6) | 0.693 (76.5)
  Cycle 2 Day 8: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 2 Day 8 | 0.0306 (14.3) | 0.0846 (19.3) | 0.0662 (68.0) | 0.214 (51.4) | 0.196 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.
  Cycle 2 Day 15 | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0435 (8.1) | 0.0266 (96.3) | 0.164 (30.7) | 0.149 (45.0)
  Cycle 3 Day 1: Predose: number analyzed (Participants) | 3 | 3 | 1 | 3 | 0
  Cycle 3 Day 1: Predose | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0120 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.144 (49.1) |
  Cycle 3 Day 1: 30 min Postdose: number analyzed (Participants) | 3 | 3 | 1 | 3 | 0
  Cycle 3 Day 1: 30 min Postdose | 0.132 (20.5) | 0.327 (33.4) | 0.716 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 1.09 (10.3) |
  Cycle 3 Day 8: number analyzed (Participants) | 2 | 3 | 1 | 3 | 0
  Cycle 3 Day 8 | 0.0314 (0.7) | 0.0785 (16.4) | 0.102 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.236 (41.1) |
  Cycle 3 Day 15: number analyzed (Participants) | 3 | 3 | 0 | 3 | 0
  Cycle 3 Day 15 | 0.0120 (NA) — Since majority of the values were LTR and data was evaluable only for 1 participant, geometric co-efficient of variation was not evaluable. | 0.0510 (14.4) |  | 0.181 (40.1) |
  Cycle 4 Day 1: Predose: number analyzed (Participants) | 2 | 3 | 0 | 1 | 0
  Cycle 4 Day 1: Predose | 0.0120 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0120 (23.9) |  | 0.0938 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 1: 30 min Postdose: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 1: 30 min Postdose | 0.0570 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.338 (23.9) |  | 0.633 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 8: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 8 | 0.0316 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.108 (19.1) |  | 0.149 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Cycle 4 Day 15: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 15 | 0.0120 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. | 0.0574 (17.3) |  | 0.0906 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable. |
  Study Drug Discontinuation Visit: number analyzed (Participants) | 2 | 2 | 3 | 2 | 1
  Study Drug Discontinuation Visit | 0.0226 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0452 (56.1) | 0.0249 (71.8) | 0.0120 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not evaluable. | 0.0374 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.

9. Secondary Outcome: Number of Participants With Objective Response Assessed According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Objective response was defined as a complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to RECIST v1.1. CR, defined as disappearance of all target lesions. PR, defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. OR=CR+PR.
Time Frame: From start of treatment until confirmation of CR or PR (up to approximately 39 months)
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
Participants
  Complete Response (CR) | 0 | 1 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Duration of Response (DoR) Assessed According to RECIST v1.1
Description: DOR was defined as the time from the first occurrence of a documented objective response to disease progression (PD) or death from any cause, whichever occurred first, as determined by the investigator according to RECIST v1.1. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: From the initial CR or PR to the time of PD or death, whichever occurs first (up to approximately 39 months)
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication. DoR was only evaluated in participants who achieved an objective response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
months |  | NA [NA to NA] — Since only one participant showed response, median and 95% confidence interval (CI) were not evaluable. |  |  |

11. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) to DHES0815A
Description: Number of participants with treatment induced and treatment-enhanced ADA are reported here. Participants were considered to have treatment-induced ADA responses if they were ADA negative at baseline and developed an ADA response following DHES0815A administration. Participants were considered to have treatment-enhanced ADA if they were ADA positive at baseline and the titer of one or more postbaseline samples is at least 4-fold greater than baseline titer (i.e., ≥ 0.60 titer units) following study drug administration.
Time Frame: Pre-dose on Day 1 of Cycles 1-4 and 42 days after last infusion (up to approximately 39 months)
Population: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
Participants
  Baseline: ADA Positive | 1 | 0 | 0 | 0 | 1
  Post-baseline: Treatment-induced ADA Positive | 0 | 1 | 1 | 0 | 0
  Post-baseline: Treatment-enhanced ADA Positive | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 to end of study (up to approximately 39 months)
Description: Safety evaluable population included all enrolled participants who received at least one dose of study medication.
Arm/Group | Dose Escalation Cohort: DHES0815A 0.6 mg/kg | Dose Escalation Cohort: DHES0815A 1.2 mg/kg | Dose Escalation Cohort: DHES0815A 2.4 mg/kg | Dose Escalation Cohort: DHES0815A 4 mg/kg | Dose Escalation Cohort: DHES0815A 6 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Cohort: DHES0815A 0.6 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 1.2 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 2.4 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 4 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 6 mg/kg (N=2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Cohort: DHES0815A 0.6 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 1.2 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 2.4 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 4 mg/kg (N=3) | Dose Escalation Cohort: DHES0815A 6 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03451162/Prot_SAP_000.pdf